# A Double-Blind, Placebo-Controlled Study of Memantine in Body focused Repetitive Behaviors

IRB20-1992 **Version: 05** 

Jon E. Grant, J.D., M.D., M.P.H. University of Chicago Chicago, IL

June 8, 2021

NCT04792645

# A Double-Blind, Placebo-Controlled Study of Memantine in Body Focused Repetitive Behavior Disorders

This clinical trial will be conducted in the spirit of Good Clinical Practice and in accordance with this IRB approved protocol. No deviation from the protocol will be implemented without the prior review and approval of the IRB except where it may be necessary to eliminate an immediate hazard to a research subject. In such a case, the deviation will be reported to the IRB as soon as possible.

#### **Investigational Agent and Dosing**

Memantine 10mg to 20mg po qday

# **Population**

The population to be studied for this trial is 100 men and women ages ≥18 years who have a current DSM-5 diagnosis of trichotillomania or skin picking disorder (i.e. a body focused repetitive behavior (BFRB)).

# **Project Goals**

The goal of the proposed study is to evaluate the efficacy and safety of memantine in 100 subjects with DSM-5 trichotillomania or skin picking disorder. Subjects will receive 8 weeks of double-blind memantine or placebo. The hypothesis to be tested is that memantine will be effective and well tolerated in patients with BFRBs compared to placebo. The proposed study will provide needed data on the treatment of disabling disorders that currently lack a clearly effective treatment.

# **Background**

Hair pulling disorder (i.e. trichotillomania) and skin picking disorder are often categorized under the umbrella term of body focused repetitive behaviors (BFRB) disorders. These repetitive, intentionally performed behaviors often cause noticeable cosmetic issues and may result in clinically significant distress or functional impairment (1-3). Although discussed in the medical literature for over one hundred years, and affecting all strata of society, there are no clear treatment approaches for people with these disorders (4). Behavioral therapy is generally regarded as the first-line treatment but trained therapists are difficult to find. In addition, there is no medication currently approved by the Food and Drug Administration for these disorders.

It appears that trichotillomania and skin picking disorder may in fact share a common neurobiology which involves an excess of activation in the mesocorticolimbic area and a lack of top-down cortical control governing response suppression. The potential effectiveness of memantine in BFRBs may be via its antagonism of the NMDA receptors in the striatum (5-6) and its potential to improve aspects of cognition by modulating glutamatergic neurotransmission in the cortex.

Recent studies using diffusion tensor imaging demonstrated that both trichotillomania and skin picking subjects exhibited significantly reduced fractional anisotropy in anterior cingulate, pre-supplementary motor area, and temporal cortices (7-8). These data suggest that the disorganization of white matter tracts in motor habit generation and suppression may underlie the pathophysiology of these disorders (7-8). Neurochemically, motor habits may rely partially on the glutamate systems. Glutamatergic dysfunction has been implicated in the pathophysiology of these disorders (9-10). Pharmacotherapies, such as memantine, that target excessive glutamatergic drive may, therefore, be expected to correct the underlying pathophysiology and symptoms of BFRBs.

Given the serious personal consequences associated with trichotillomania and skin picking disorder, and the likelihood of success of memantine in treating both disorders, the aim of the present study was to examine the efficacy and safety of memantine vs placebo in adults with trichotillomania or skin picking disorder using a double-blind, placebo-controlled design.

We hypothesize that memantine will be more effective than placebo in reducing the frequency of hair pulling and skin picking and in improving overall psychosocial functioning after 8 weeks of treatment when compared to baseline.

# **Primary Aim/Objective**

The aim of the present study is to examine the efficacy and safety of memantine vs placebo in adults with trichotillomania and skin picking disorder.

Primary Endpoint(s):

The primary efficacy measure will be the change in hair pulling or skin picking frequency and urges to pull hair or pick skin for the past week as indicated by change in total score on the *NIMH Symptom Severity Scale* (for TTM or Skin Picking)(11). The primary efficacy end points will be the change in these measures from baseline to week 8.

# **Secondary Aim/Objective**

A secondary aim of the study is to examine the effects of memantine vs placebo on self-report measures of hair pulling, skin picking, quality of life, and measures of mood and anxiety.

Secondary Endpoint(s):

Secondary efficacy measures include the change in number of days per week pulling/picking, the Clinical Global Impressions—Improvement Scale (CGI-I) rated global improvement of symptoms over time (results will be dichotomized as improved [CGI-I ratings of 1 or 2 very much/much improved] or not improved [CGI-I ratings of 3-7]) (12), the self-report Massachusetts General Hospital Hairpulling Scale (13), the Skin Picking Symptom Assessment Scale (14), the Quality of Life Inventory (15), the Sheehan Disability Scale (16), the Hamilton Depression Rating Scale (17), the Hamilton Anxiety Rating Scale (18), the Tridimensional Personality Questionnaire (19), the Autism Spectrum Quotient (20), and the Barratt Impulsiveness Scale (21).

# Methodology

100 individuals with trichotillomania or skin picking disorder will be recruited for a double-blind, placebo-controlled pilot study in which memantine or placebo is administered in a 1:1 fashion. All 100 subjects will have trichotillomania or skin picking disorder per DSM-5 criteria. Following baseline measures, all subjects will be randomized to either memantine or placebo and seen every 2 weeks for the 8-week study period.

Participants will be started at 10mg po qday for 2 weeks, then 20mg po qday for the remaining 6 weeks. Participants will only go up to the full dose if clinically needed. Efficacy and safety measures will be performed at each visit.

The study will be conducted in accordance with the International Conference on Harmonization Guideline for Good Clinical Practice, all local ethical and legal requirements, and the World Medical Assembly (Declaration of Helsinki). The study protocol and procedures will be approved by the University of Chicago's institutional review board prior to any recruitment. Written informed consent will be required for study participation.

Randomization of drug will be conducted in blocks of eight, with 4 subjects in the memantine arm and 4 subjects in the placebo arm. In event of an emergency, the blind will be assessable to the study subject by calling the pharmacy number listed on the medication bottle. In this event, the study subject will be discontinued from the medication, and a safety follow-up visit will be scheduled one week following discontinuation. The study subject will not know what arm of the study they are on otherwise. The investigational pharmacy will follow proper accountability procedures in regards to both randomization of the study drug and holding of the blind.

## **Subjects:**

#### Inclusion criteria:

- 1) men and women age ≥18 years;
- 2) current DSM-5 trichotillomania or skin picking disorder; and
- 3) Ability to understand and sign the consent form.

#### Exclusion criteria:

- 1) Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
- 2) Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
- 3) Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
- 4) Past 12-month DSM-5 diagnosis of psychosis, bipolar disorder, mania, or a substance or alcohol use disorder
- 5) Illegal substance use based on urine toxicology screening
- 6) Stable dose of medications for at least the past 3 months
- 7) Previous treatment with memantine

8) Cognitive impairment that interferes with the capacity to understand and selfadminister medication or provide written informed consent

#### **Baseline Assessments:**

Those subjects who appear appropriate for the study, based on telephone screening, will be invited for a baseline assessment. The duration of the baseline assessment will be approximately 90 minutes and will include the following: informed consent, demographic data, concomitant medications, and family history data. There will also be a physical examination (including weight, and vital signs, urine pregnancy test for women of childbearing years and urine drug screen). Finally, the subjects will undergo a psychiatric evaluation (using the MINI International Neuropsychiatric Interview).

In addition, the following instruments will be completed at the screening visit: 1) NIMH Trichotillomania Symptom Severity Scale (or the same scale modified for skin picking); 2) Sheehan Disability Scale; 3) Massachusetts General Hospital Hairpulling Scale; 4) the 17-item Hamilton Rating Scale for Depression (HAM-D); 5) the 17-item Hamilton Rating Scale for Anxiety (HAM-A); 6) Clinical Global Impression (Improvement and Severity) scale; 7) Cambridge Caffeine Use Questionnaire; 8) The Dietary Fat and Free Sugar Questionnaire and 9) the Quality of Life Inventory; 10) Cambridge-Chicago Trait Scale (12); 11) the Skin Picking Symptom Assessment Scale (SP-SAS); 12) the Autism Spectrum Quotient (AQ-10); and the Barratt Impulsiveness Scale (BIS). In addition, subjects will undergo cognitive assessments at baseline and study endpoint.

**Cognitive Assessments:** Assessments of cognitive control will be comprised of several valid paradigms (See below). These tasks are designed to probe dissociable neural circuitry and cognitive processes likely to be implicated in the pathophysiology of addictions. Task order was chosen arbitrarily and will be applied consistently across subjects, to minimize possible confounding factors of differences in task order across participants.

The following tasks will be administered at baseline and final visits:

- -Stop Signal Task of Inhibitory Control (SST)
- -Intra-dimensional/Extra-dimensional Set Shift Task (ID/ED task)
- -One Touch Stockings Task (OTS)
- -Rapid Visual Processing Task (RVP)
- -Spatial Working Memory Task (SWM)
- -Cambridge Gambling Task (CGT)

#### **Following-Up Visit Assessments**

All follow-up visits will include all psychiatric measures (except the MINI which will be done at baseline only) and safety measures (adverse events, vital signs, C-SSRS). There will be four follow up visits for a total of five visits.

## **Subject Compensation**

Subjects will be compensated \$20 per visit, for a total of \$100. Compensation will be given in the form of a check at the end of the study, as per University of Chicago protocol.

#### **Safety Assessments**

Safety and tolerability will be assessed using spontaneously reported adverse events data, Columbia–Suicide Severity Rating Scale (C-SSRS), vital signs, and by evaluating premature

termination. Safety assessments (C-SSRS, sitting blood pressure, heart rate, adverse effects, and concomitant medications) will be documented at each visit. Subjects who are an immediate suicide risk will be removed from the study and appropriate clinical intervention (e.g. hospitalization) will be arranged. Urine pregnancy tests will be performed at the initial visit. Subjects who have a positive urine pregnancy test will be excluded from the study. Assessment of side effects will be done at each visit. AEs will be coded by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (Med-DRA) Version11.1. The incidences of all AEs will be summarized descriptively. In terms of vital signs, those subjects with abnormal blood pressures will be assessed for symptoms of hypo- or hypertension. Asymptomatic subjects will be evaluated each visit for changes in vital signs. In the case of hypertensive emergencies (BP greater than 210/120), appropriate referral to the emergency room will be made. In the case of hypotension (BP less than 90/60), participants will be evaluated for symptoms of hypotension and if symptomatic, appropriate interventions will be made.

## **Subject Withdrawal**

If a subject withdraws from the study, all instruments administered at the screening visit will be completed at the final visit. These will be conducted when the subject is able to come in for an early termination visit. Withdrawn subjects will be given the phone number of the principal investigator as well as the phone numbers of local resources for trichotillomania and skin picking.

## **Data and Safety Monitoring Plan**

- 1. Responsibility for Data and Safety Monitoring
  The PI will have overall responsibility for monitoring the integrity of study data and participant safety.
- 2. Procedures for Monitoring Participant Safety
  The PI will implement the following procedures to ensure data integrity and the safety of participants during the study.
  - A number of elements of the research plan are intended to minimize the risks of study participation. If subjects become actively suicidal with intent and plan to kill themselves, the PI will evaluate them and refer them for immediate non-study treatment. Any participant endorsing suicidal thoughts with intent and plan will be immediately evaluated by the PI and referred to a higher level of care if clinically indicated.
  - The PI will evaluate patient safety and resolve any safety issues if necessary, as such issues arise. The PI will also be responsible for preparing written summary reports of adverse events and will prepare a written report summarizing any decisions that are made pertaining to participant disposition.
  - Data integrity and confidentiality will be safeguarded as discussed above in the Data Management and Statistical Analysis section under Research Methods.

## **Monitoring Committee**

We will establish a monitoring committee and define in detail its role, its composition, and its operating procedures for reviewing patient safety and data from this study. The monitoring committee, comprised of three individuals independent of personnel involved in the study,

including a psychiatrists and a statistician, will come together via conference call yearly. The committee will use a standardized approach employing contemporary bio statistical, psychiatric/psychological, and ethical principles to review study design and interim data every year. The committee will audit the records from the study and will ensure the data are being collected, managed and protected. The committee will have the ability to ask for more frequent reviews at any time if they deem it necessary. In addition, the PI will inform the committee of any serious adverse event.

The PI will prepare a specific report for the committee in advance of each meeting. Attention will be given to data quality and timeliness, recruitment, risk versus benefit, adverse events and other factors that could affect study outcome.

## 3. Reporting Adverse Events

- Any serious adverse event will be reported to the Institutional Review Board (IRB) at the University of Chicago in a full written report within 10 working days of the event. For fatal/life-threatening serious adverse events, the PI will notify the IRB Chair by phone immediately.
- Any moderate adverse event which appears definitely, probably, or possibly related to study participation will be reported to the University of Chicago IRB in writing within 20 working days.
- Any mild adverse event will be summarized in the IRB annual progress reports.

#### **Statistical Analysis**

## Design/Randomization

The study is a double-blind, placebo-controlled study. Participants will be randomized (1:1) to receive memantine or placebo by the University of Chicago Investigational pharmacy in block sizes of eight, using computer-generated randomization with no clinical information.

Due to the pandemic of COVID19, study participants can perform their baseline and follow-up visits online using encrypted Zoom instead of in person visits. All inventories will be assessed. Blood samples and urine toxicology, however, will be at the discretion of the study PI. In cases where they are considered medically necessary, the participant can have them drawn locally and submitted to the study team.

#### **Efficacy Analysis**

For statistical analysis, the full-analysis set will be defined as all participants who took at least 1 dose of the study drug and had at least 1 post-randomization primary efficacy assessment. The safety-analysis set will be defined as all randomized participants who took at least 1 dose of the study drug and completed at least 1 post-randomization safety assessment. Participants with trichotillomania and skin picking disorder will be grouped as one BFRB group.

We will compare the baseline characteristics of both groups using Fisher's exact test for categorical variables and the t test for continuous variables. We will calculate adherence to treatment, based on the number of pills returned at each visit, as the number of pills taken divided by the number of days in the study  $\times$  100%.

# Primary endpoint analysis

The primary outcome measure will be the change from first randomization visit to study endpoint in total composite score on the NIMH Trichotillomania/Skin Picking Symptom Severity Scale.

The primary analysis of efficacy for continuous measures will be analysis of variance (ANOVA), with terms for treatment to assess differences between treatment groups in the change from first randomization visit to endpoint using the last observation carried forward. The primary analysis for global improvement and response categories will be the Cochran-Mantel-Haenszel test using the last observation carried forward. The primary analysis for ≥5% reduction in weight will be Fisher's exact test using the last observation carried forward.

# Secondary endpoints analyses

Secondary outcome measures will include the change from first randomization visit to study endpoint in CGI severity and improvement scales, self-reported hair pulling behavior using the MGH-HPS, self-reported skin picking behavior using the SP-SAS, the change in depressive and anxiety symptoms, change in quality of life, and impacts on personality markers. We will use a longitudinal analysis comparing the rate of change of the outcome during the treatment period between groups. The difference in rate of change will be estimated by random regression methods. The model for the mean of the outcome will include terms for treatment, time, and treatment-by-time interaction. To account for the correlation of observations within participants, we will use SAS procedure MIXED with a first-order antedependence covariance structure. The longitudinal analyses will use all available observations from all time points from all participants who completed a randomization visit evaluation.

## Safety analyses

We will evaluate differences between groups in the incidence of treatment-emergent adverse events using Fisher's exact test. Descriptive statistics will be used to evaluate changes in laboratory values, blood pressure and heart rate.

# Sample Size

The sample size was calculated for the primary endpoint of change from randomization. For 80% power to compare the change from randomization, assuming a true effect size of 0.5 between treatment group and the placebo group, 30 participants with a BFRB will be needed in each treatment group based on a 2-group t test at the .05 level of significance. Given the low rates of adverse events expected with memantine, we expect few drop-outs from the study.

# **Data Management Plan**

Data collected will consist of demographic data, subjective (self-report questionnaires, interview responses, ratings), and physiological (weight, heart rate and blood pressure). Access to individually identifiable private information about human subjects will be limited to Dr. Grant and their staff and will be collected specifically for the proposed research project. All collected data will be stored utilizing a 4-digit subject identification code, linked to separately stored identifying information via a coded log only available to the PI.

The gender ratio of trichotillomania and skin picking disorder have been estimated to be approximately 3:1 (female:male). We will also make every effort to include a racially/ethnically

diverse study population. The year 2010 Chicago census is 2,695,598 (US Census Bureau, 2011). The year 2010 Chicago race distribution is as follows: white 47.1%, African/African-American 33.9%, Asian/Asian-American 6.2%, Native American 1.0%, or other race/not identified (11.8%). A total of 28.9% of the population also identified as Hispanic/Latino allowing for a diverse population sample (year 2010, US Census Bureau, Chicago, IL). We will make every effort to ensure that members of both genders and diverse racial, ethnic, and socioeconomic groups are adequately represented in the proposed study.

The PI will implement the following procedures to ensure data integrity and the safety of participants during the study: A number of elements of the research plan are intended to minimize the risks of study participation. For example, the study exclusion criteria exclude patients who are experiencing clinically significant suicidality or require a higher level of care than outpatient. If this is indicated, the PI will evaluate them and refer them for immediate non-study treatment (for example, inpatient or additional pharmacologic treatment). The PI will carefully monitor ratings on the Columbia Suicide Severity Rating Scale and the Hamilton Depression Rating Scale; any participant endorsing suicidal thoughts, will be immediately evaluated by the PI and referred to a higher level of care if clinically indicated. The PI will evaluate patient safety at each visit and resolve any safety issues more frequently if necessary, as such issues arise. The PI will also be responsible for preparing written summary reports of adverse events and will prepare a written report summarizing any decisions that are made pertaining to participant disposition.

#### **Ethical Considerations**

This study will be conducted according to US and international standards of Good Clinical Practice (FDA regulations 21 CFR 312 for IND studies and FDA guidance E6) for all studies. Applicable government regulations and University of Chicago research policies and procedures will also be followed.

This protocol and any amendments will be submitted to the University of Chicago Institutional Review Board (IRB) for formal approval to conduct the study. The decision of the IRB concerning the conduct of the study will be made in writing to the investigator.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB. The formal consent of a subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. This consent form must be signed by the subject and the investigator-designated research professional obtaining the consent.

#### REFERENCES

- 1. Grant JE, Chamberlain SR. Trichotillomania. Am J Psychiatry. 2016 Sep 1;173(9):868-74. doi: 10.1176/appi.ajp.2016.15111432. PMID: 27581696; PMCID: PMC5328413.
- 2. Woods DW, Flessner CA, Franklin ME, et al. The Trichotillomania Impact Project (TIP): exploring phenomenology, functional impairment, and treatment utilization. J Clin Psychiatry. 2006;67:1877–1888
- 3. Grant JE, Odlaug BL, Chamberlain SR, Keuthen NJ, Lochner C, Stein DJ. Skin picking disorder. Am J Psychiatry. 2012 Nov;169(11):1143-9. doi: 10.1176/appi.ajp.2012.12040508. PMID: 23128921.
- 4. Bloch MH, Landeros-Weisenberger A, Dombrowski P, et al. Systematic review: pharmacological and behavioral treatment for trichotillomania. Biol Psychiatry. 2007;62:839–846.
- 5. Krystal JH, Petrakis IL, Krupitsky E, Schutz C, Trevisan L, D'Souza DC. NMDA receptor antagonism and the ethanol intoxication signal: from alcoholism risk to pharmacotherapy. Ann N Y Acad Sci. 2003;1003:176–184
- 6. Ma YY, Cepeda C, Cui CL. The role of NMDA receptors in drug addiction. Int Rev Neurobiol. 2009;89:131–146
- 7. Chamberlain SR, Hampshire A, Menzies LA, Garyfallidis E, Grant JE, Odlaug BL, Craig K, Fineberg N, Sahakian BJ (2010) Reduced brain white matter integrity in trichotillomania: a diffusion tensor imaging study. Arch Gen Psychiatry 67:965–971.
- 8. Grant JE, Odlaug BL, Hampshire A, Schreiber LR, Chamberlain SR. White matter abnormalities in skin picking disorder: a diffusion tensor imaging study. Neuropsychopharmacology. 2013 Apr;38(5):763-9. doi: 10.1038/npp.2012.241. Epub 2012 Nov 29. PMID: 23303052; PMCID: PMC3671993.
- 9. Grant JE, Oldaug BL, Kim SW. 2009. A double-blind, placebo-controlled trial of a glutamate modulating agent, N-acetyl cysteine, in the treatment of trichotillomania. Arch Gen Psychiatry 66(7): 756-763
- 10. Grant JE, Chamberlain SR, Redden SA, Leppink EW, Odlaug BL, Kim SW. N-Acetylcysteine in the Treatment of Excoriation Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):490-6. doi: 10.1001/jamapsychiatry.2016.0060. PMID: 27007062.
- 11. Swedo SE, Leonard HL, Rapoport JL, et al: A double-blind comparison of clomipramine and desipramine in the treatment of trichotillomania. New England Journal of Medicine 321:497-501, 1989
- 12. Guy W: ECDEU Assessment Manual for Psychopharmacology. US Dept Health, Education and Welfare publication (ADM) 76-338. Rockville, MD: National Institute of Mental Health, 218-222, 1976.
- 13. Keuthen NJ, O'Sullivan RL, Ricciardi JN, et al: The Massachusetts General Hospital (MGH) Hairpulling Scale, 1: development and factor analysis. Psychotherapy and Psychosomatics 64:141-145, 1995
- 14. Grant JE, Odlaug BL, Chamberlain SR, Kim SW. A double-blind, placebo-controlled trial of lamotrigine for pathological skin picking: treatment efficacy and neurocognitive predictors of response. J Clin Psychopharmacol. 2010 Aug;30(4):396-403. doi: 10.1097/JCP.0b013e3181e617a1. PMID: 20531220; PMCID: PMC3172612.

- 15. Frisch MB, Cornell J, Villaneuva M: Clinical validation of the Quality of Life Inventory: a measure of life satisfaction for use in treatment planning and outcome assessment. Psychological Assessments 4:92-101, 1993
- 16. Sheehan DV. The Anxiety Disease. New York: Scribner's, 1983
- 17. Hamilton, M: A rating scale for depression. Journal of Neurosurgery & Psychiatry 23:56-62, 1960
- 18. Hamilton, M: The assessment of anxiety states by rating. British Journal of Medical Psychology 32:50-55, 1959
- 19. Cloninger CR, Przybeck TR, Svrakic DM. The Tridimensional Personality Questionnaire: U.S. normative data. Psychol Rep. 1991 Dec;69(3 Pt 1):1047-57. doi: 10.2466/pr0.1991.69.3.1047. PMID: 1784653.
- 20. Allison C, Auyeung B, Baron-Cohen S. Toward brief "red flags" for autism screening: the short autism spectrum quotient and the short quantitative checklist in 1,000 cases and 3,000 controls. Journal of the American Academy of Child and Adolescent Psychiatry 51(2):202-12, 2012.21.
- 21. Barratt E: Anxiety and impulsiveness related to psychomotor efficiency. Percept Mot Skills 1959; 9:191–198.